CLINICAL TRIAL: NCT02134743
Title: Evaluation of the Stability of Implants With Two Different Surface Treatments: a Randomized Clinical Trial
Brief Title: Evaluation of the Stability of Implants With Two Different Surface Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Michele Novellino, PHD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 18911913.7.0000.0075
Record Dates: First submitted 2014-05-04; First posted 2014-05-09 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Dental Implant Failed; Pre-osseointegration Failure of Dental Implant
Keywords: dental implant; Surface energy; Hydrophilicity; Contact angle; Titanium implant roughness; Surface conditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): At this group the patients will receive dental implants which have a modified SLA surface. These surface have wettability, which could improve and accelerate the osseointegration.Intervention: implant placement.
  Interventions: Procedure: Implant surgery
- Control Group (Active Comparator): The patient of this group will receive implant with conventional surface, SLA (Sandblasted and Acid-Etched Surface).Intervention: implant placement.
  Interventions: Procedure: Implant surgery

INTERVENTIONS:
Procedure: Implant surgery — Dental implant surgery with two different kinds of implant surface (SLA and modified SLA)
  Other Names: Neodent Neoporos (SLA surface); Neodent Acqua (Modified SLA surface)

SUMMARY:
The aim of this study is to compare the stability of dental implant surface treated by sandblasting abrasive particles and acid subtraction (Control) with hydrophilic surfaces dental implants (chemical) and with a higher surface energy (Test) for a period of 16 weeks after installation. The evaluation will be made by analyzing the resonance frequency (Ostell). The hypothesis to be tested will be that implants with hydrophilic surface show increased secondary stability prior to the implants treated by acid etching.

DETAILED DESCRIPTION:
The selected patients will be randomly divided into two groups by computer-generated list. The control group will receive implant surface treated by acid etching and test group receive implants with hydrophilic surface (Test). Both the test and the control group will undergo the same pre-surgical, surgical and post-surgical protocols.

The evaluation of the implant will be done by the analysis of resonant frequency wich will be performed on each implant with Osstell (Integration Diagnostics AB, Goteborg, Sweden) immediately after implant placement (baseline) and at follow-up sessions (1st, 2nd, 3rd, 5th, 8th, 12th and 16th weeks after installation) and coefficient of implant stability (ISQ) on these dates will be measured on a scale from 0 to 100. The smartpeg be used with special developed Healing without the use of pillars or intermediaries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had lost teeth in the posterior maxilla (region of premolars and molars, can be interspace or free end) in need of restoration with implant-supported prostheses
* Able to understand and sign a waiver of informed free consent
* Good oral hygiene
* The receiving implant sites must have at least 3 months of healing after tooth extraction, proper height and width to install an implant of 4.3 mm in diameter and 10 mm of high.

Exclusion Criteria:

* Patients requiring implants in the mandible or anterior maxilla (bone type I and II), or to submit any of the following conditions: general contraindications for surgical procedures, uncontrolled diabetes, severe bruxism or clenching, pregnant and lactating women, active periodontal disease, smoking and use of alcohol or drugs
* Patients who underwent radiotherapy near the buccal cavity regions chemotherapy and those who use or have recently used bisphosphonates, such as alendronate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Loss of implant | 4 months after surgery
  If the implant has been not integrated to the bone!

SECONDARY OUTCOMES:
Implant stability (ISQ) | Baseline, 1 to 16 weeks (4 months)
  If the implant get successively and it has been integrated to bone. The stability will be evaluated at the surgery day (T0), one week after surgery (T1),after 2 weeks (T2), after 3 weeks (T3), after 5 weeks (T4), after 8 weeks (T5), after 12 weeks (T6) and after 16 weeks (T7).

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry School - University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Bornstein MM, Wittneben JG, Bragger U, Buser D. Early loading at 21 days of non-submerged titanium implants with a chemically modified sandblasted and acid-etched surface: 3-year results of a prospective study in the posterior mandible. J Periodontol. 2010 Jun;81(6):809-18. doi: 10.1902/jop.2010.090727. PMID 20450357
- [Background] Schwarz F, Wieland M, Schwartz Z, Zhao G, Rupp F, Geis-Gerstorfer J, Schedle A, Broggini N, Bornstein MM, Buser D, Ferguson SJ, Becker J, Boyan BD, Cochran DL. Potential of chemically modified hydrophilic surface characteristics to support tissue integration of titanium dental implants. J Biomed Mater Res B Appl Biomater. 2009 Feb;88(2):544-57. doi: 10.1002/jbm.b.31233. PMID 18837448
- [Result] Degidi M, Piattelli A, Shibli JA, Perrotti V, Iezzi G. Bone formation around one-stage implants with a modified sandblasted and acid-etched surface: human histologic results at 4 weeks. Int J Periodontics Restorative Dent. 2009 Dec;29(6):607-13. PMID 20072738